CLINICAL TRIAL: NCT00916994
Title: One-arm, International, Multi-center With Competitive Recruitment, Prospective Study to Assess the Safety and Efficacy of OrthoSpace's InSpace™ in Rotator Cuff Tear Subjects Scheduled for Surgery of the Rotator Cuff
Brief Title: Prospective Study for Safety and Efficacy of InSpace™ in Rotator Cuff Tear Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OrthoSpace Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP-04
Record Dates: First submitted 2009-06-07; First posted 2009-06-10 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2013-06

CONDITIONS: Rotator Cuff Tear
Keywords: Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SpaceGuard Balloon implantation (Experimental)
  Interventions: Device: SpaceGuard Balloon

INTERVENTIONS:
Device: SpaceGuard Balloon — Positioning of the balloon into the subacromial space between the humerus head and the acromion

SUMMARY:
Title: One-arm, international, multi-center with competitive recruitment, prospective study to assess the safety and efficacy of OrthoSpace's InSpace™ in rotator cuff tear subjects scheduled for surgery of the rotator cuff - A pivotal study

Device: OrthoSpace's Biodegradable Implanted Balloon (InSpace)

Study population: Rotator Cuff tear subjects scheduled for arthroscopy.

Number of subjects: Up to 70 subject for data analysis.

Number of sites: At least 4 sites in Israel.

Main Inclusion criteria: Informed consent, diagnosed with Rotator Cuff tear.

Main Exclusion criteria: Former surgery on affected shoulder, sever illness, significant shoulder co morbidities.

Follow up period: 12 months. Visits at hospital before discharge at 1-2 days post implantation, 7-10 days post implantation, 3 weeks post implantation, 6 weeks post implantation, 3,6 and 12 months post implantation.

Primary goal: To assess the safety of the SpaceGuard in Rotator Cuff tear subjects.

Secondary goals: To assess the effectiveness of the SpaceGuard in the study population. The effectiveness will be assessed by terms of good positioning of the SpaceGuard and subsequent follow-up non migration, surgeon satisfaction, pain relief and time to pain relief, Range of Motion (ROM) and time to ROM with the SpaceGuard.

Primary end point: Serious Adverse Event rate related to the device and/or system complication.

Secondary end points: Surgeon dissatisfaction following the deployment of SpaceGuard, migration of the balloon shown by ultrasound/ X-ray/MRI at relevant follow-up visits, lost of ROM and pain enhancement.

DETAILED DESCRIPTION:
The OrthoSpace's InSpace™ biodegradable sub-acromial spacer (balloon) will be inserted at the end of the routine arthroscopy between the humerus head and the acromion.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older.
2. Diagnosed with Rotator Cuff tear and are scheduled for surgery.
3. X-Ray of treated shoulder with no unrelated pathology and imaging (ultrasound or MRI) showing Rotator Cuff tear.
4. Persistent pain and functional disability for at least 4 months.
5. Documented failure of conservative treatment.
6. Blood work up to two weeks before implantation as follow:

   * Normal CBC
   * Normal electrolytes (potassium, chloride, phosphorous, sodium)
   * Absolute neutrophil count (ANC) ≥ 1,800 cells/mm3
   * Platelets ≥ 100,000 cells/mm3
   * Hemoglobin ≥ 10.0 g/dl
   * Adequate renal function, with serum creatinine ≤ 2.0 mg/dl
   * Adequate liver function, with serum bilirubin < 2.0 mg/dl
   * Adequate liver function with SGOT/SGPT < 2.5 x the upper normal limit
   * Normal values of the PT, PTT and INR tests
7. Negative for HIV and Hepatitis B or C
8. Mentally and physically able to fully comply with this protocol including adhering to follow-up schedule and requirements
9. For Woman of Child Bearing Potential (WOCBP), negative pregnancy test and willingness to use birth control during the study.
10. Singed Informed Consent Form.

Exclusion Criteria:

1. Evidence of significant osteoarthritis or cartilage damage in the shoulder.
2. Evidence of glenohumeral instability.
3. Previous surgeries of the shoulder .
4. Evidence of major joint trauma, infection, or necrosis in the shoulder.
5. Patients unable to provide informed consent due to language barrier or mental status.
6. Patients with a major medical condition that would affect quality of life and influence the results of the study (Including, but not limited to HIV, hepatitis, active malignancy in the past 5 years, transmural MI, CVA and other impaired neurological status, CHF or unstable angina in the past 6 months).
7. Patients unwilling to be followed for the duration of the study.
8. Acute infection requiring intravenous antibiotics at the time of screening.
9. Other shoulder pain of unknown etiology.
10. Paget's disease, osteomalacia or any other metabolic bone disease.
11. Severe diabetes mellitus requiring daily insulin management.
12. Bleeding disorders.
13. Known cognitive disorder.
14. Concurrent participation in any other clinical study.
15. Physician objection.
16. Subjects with sign of cervical root irritation.
17. Chronic lung disease
18. Trauma subjects
19. For WOCBP, a positive pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-07; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The study's primary goal is to assess the safety of the SpaceGuard and implantation procedure, in the study population. Safety of the SpaceGuard will be assessed by reporting system related adverse events. | 12-36 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Eliyahu Adar, MD, Principal Investigator — Wolfson Medical Center
Locations (1):
- Wolfson Medical Center, Holon, Israel